CLINICAL TRIAL: NCT03859492
Title: Screening Contrast Enhanced Mammography (CEDM) in Intermediate and High-Risk Patient Populations
Brief Title: Screening CEDM in Intermediate and High-Risk Patient Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bhavika Patel, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18-010602; NCI-2022-11058 (Registry Identifier: NCI)
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are prospectively assigned to the CEDM /screening intervention which may lead to additional screening or biopsy based on the study schema.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermediate or high-risk breast cancer subjects (Experimental): Subjects with a negative mammogram who are intermediate or high-risk for breast cancer will get supplemental screening with contrast enhanced digital mammography (CEDM)
  Interventions: Device: Contrast Enhanced Digital Mammography

INTERVENTIONS:
Device: Contrast Enhanced Digital Mammography — High-resolution, low-energy, full-field digital mammography (FFDM) image and contrast-enhanced image
  Other Names: CEDM

SUMMARY:
This research study is being done to determine if Contrast Enhanced Digital Mammography (CEDM) can improve breast cancer detection and can be used as an additional screening method to the standard mammographic screening.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 35 and had a negative routine mammogram within 6 months.
* Qualifies as intermediate or high-risk (>15% lifetime risk of breast cancer as defined by IBIS version 8).

Exclusion Criteria:

* Known breast cancer
* Previously had negative MBI or MRI within 12 months of study
* Pregnant or lactating
* Contraindication to intravenous iodinated contrast
* Unable to understand or sign informed consent
* Self-reported signs or symptoms of breast cancer

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 461 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Breast Cancer | 3 years
  Number of subjects diagnosed with breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Bhavika Patel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials